CLINICAL TRIAL: NCT01060488
Title: A Phase III, Multicentric, Open-label, Randomised, Comparative, Parallel Group Study of (GHRH + Arginine) Combination Test vs. Insulin Tolerance Test (ITT) in the Diagnosis of Adult Growth Hormone Deficiency (AGHD)
Brief Title: Comparative Validation of the Growth Hormone Releasing Hormone and Arginine Test for the Diagnosis of Adult Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Dr. Laurence Fresneau, Merck Serono s.a.s., an Affiliate of Merck KGaA, Darmstadt, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IMP24689
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2011-07

CONDITIONS: Growth Hormone Deficiency
Keywords: GH secretion tests; adverse effects; adult growth hormone deficiency; growth-hormone releasing hormone and arginine test; insulin tolerance test; GHRH + Arginine test
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: (Active Comparator)
  Interventions: Other: GHRH+Arg, GHRH+Arg, ITT
- Group 2: (Active Comparator)
  Interventions: Other: ITT, ITT, GHRH+Arg.

INTERVENTIONS:
Other: GHRH+Arg, GHRH+Arg, ITT — GHRH+Arg repeatability test (2 tests) + comparison with one IT test
  Arms: Group 1:
Other: ITT, ITT, GHRH+Arg. — IT repeatability test (2 tests) + comparison with one GHRH+Arg test
  Arms: Group 2:

SUMMARY:
The aim of the study is to determine the specificity and sensitivity of the combined growth hormone releasing hormone (GHRH) + Arginine test in healthy volunteers, subjects with highly probable adult growth hormone deficiency (AGHD) and subjects who were probably free of AGHD.

DETAILED DESCRIPTION:
The randomisation was carried out before the first test was performed. In order to be informed of the subject's randomisation group, the investigator phoned the access number given to him/her. The subject's allocation to a given randomisation arm was determined on the basis of a centralised randomisation (answering service), balanced per group of subjects with a minimisation on 2 criteria: age and BMI.

This was a centralised randomisation using a Interactive Voice Response System (IVRS) which was balanced in each of the following 3 categories of subjects:

* Category A = healthy volunteers,
* Category B = subjects with a strong probability of deficit in GH,
* Category C = subjects with a low probability of deficit in GH.

In each of these 3 categories, the subjects underwent 3 tests whose sequences were determined by the following randomisation group:

* Group 1: GHRH+Arg, GHRH+Arg, ITT or
* Group 2: ITT, ITT, GHRH+Arg.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged over 18 years and under 60 years,
* Female or male,
* Subjects not treated by GH or having stopped the treatment more than 15 days ago,
* Effective contraception in women of childbearing age: hormonal contraception or use of female condom and spermicides or use of diaphragm and spermicides or Intra Uterine Device (IUD),
* Signed informed consent,
* Subjects possessing social security cover.
* Subjects having at least one of the following criteria were considered as subjects with a high probability of presenting a GH deficit:

  * Subjects with a tumour of the hypothalamo-hypophyseal region (hypophyseal adenomata, craniopharyngioma, meningioma, etc.) in whom the presence of a hypophyseal insufficiency in GH must be tested preoperatively or postoperatively, or
  * Subjects presenting a secondary ante-hypophyseal insufficiency to an inflammatory, infectious, post-traumatic pathology or to a hypophyseal necrosis, whose hypophyseal functional condition has already been documented and for whom a revaluation of GH secretion is desired, or
  * Subjects having undergone, as adults, an irradiation hypothalamo-hypophyseal region, or a suprasellar irradiation, in a clinical context of GH deficit, or
  * Subjects with a known organic ante-hypophyseal insufficiency beginning in childhood and with at least 1 associated deficit excluding prolactin.
* Subjects having at least one of the following criteria were considered as subjects with a low probability of presenting a GH deficit:

  * Subjects with known idiopathic isolated GH deficit starting in childhood and for whom a new growth hormone secretion test is desired, or
  * Subjects with non-operated microadenoma (< 1 cm of diameter), or
  * Subjects with fortuitously discovered intrasellar image (e.g. Rathke's pocket cyst).

The third category of subjects eligible was made of healthy volunteers.

Exclusion Criteria:

* Subjects presenting a coronary history or whose electrocardiographic signs evoke an ischemic pathology,
* Subjects presenting a history of cerebrovascular insufficiency,
* Subjects presenting a history of epilepsy,
* Subjects with an evolutive acromegalia or an evolutive Cushing's syndrome,
* Subjects presenting a known intolerance to arginine, GHRH or insulin,
* Hyperkalemic subjects,
* Diabetic subjects (Type 1 or Type 2),
* Very obese subjects (BMI > 40),
* Subjects presenting a severe, hepatic, renal, tumoral evolutive affection or metabolic or respiratory acidosis,
* Subjects with known immuno-depression,
* Subjects with psychiatric disorders,
* Subjects presenting Parkinson's disease or Parkinsonian syndromes treated by Levodopa®,
* Subjects treated by drugs directly affecting the hypophyseal secretion of somatotrophin (e.g. clonidine, levodopa) or provoking the release of somatostatin, antimuscarinic agents (atropine),
* Subjects with untreated hypothyroidism or subjects treated by anti-thyroid synthesis drugs,
* Participation in another biomedical research programme less than 3 months previously,
* Known evolutive pregnancy or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2004-01; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Level of GH peak (recorded following stimulation tests) | within 120 min after stimulation (blood samples were tacken at T0(before), T15, T30, T45, T60, T90 and T120 min after stimulation).

SECONDARY OUTCOMES:
It was asked to the patients to evaluate acceptability of each test via a visual analogic scale. | After each test and before leaving the hospital (the day of the test)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Chanson, MD, Professor, Principal Investigator — CHU Bicêtre, Endocrinology and Reproductive Diseases Department
Locations (1):
- CHU Bicêtre, Endocrinology and Reproductive Diseases Department, Le Kremlin-Bicêtre, France

REFERENCES:
- [Result] Chanson P, Cailleux-Bounacer A, Kuhn JM, Weryha G, Chabre O, Borson-Chazot F, Dubois S, Vincent-Dejean C, Brue T, Fedou C, Bresson JL, Demolis P, Souberbielle JC. Comparative validation of the growth hormone-releasing hormone and arginine test for the diagnosis of adult growth hormone deficiency using a growth hormone assay conforming to recent international recommendations. J Clin Endocrinol Metab. 2010 Aug;95(8):3684-92. doi: 10.1210/jc.2010-0295. Epub 2010 May 19. PMID 20484474